CLINICAL TRIAL: NCT03745053
Title: XLIMus Drug Eluting Stent: a randomIzed Controlled Trial to Assess Endothelization
Acronym: XLIMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardionovum GmbH (Industry)
Collaborators: Mediolanum Cardio Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XLIMIT
Record Dates: First submitted 2018-11-09; First posted 2018-11-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomized multi-centre controlled trial
Who Masked: Outcomes Assessor
Masking Description: The members of the Event Adjudication Committee and the Core Lab will be blinded to the patient assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XLIMUS DES (Experimental): Xlimus DES Implantation during coronary angioplasty
  Interventions: Device: Xlimus DES Implantation during coronary angioplasty
- Synergy DES (Active Comparator): Synergy DES Implantation during coronary angioplasty
  Interventions: Device: Synergy DES Implantation during coronary angioplasty

INTERVENTIONS:
Device: Xlimus DES Implantation during coronary angioplasty — Xlimus DES Implantation during coronary angioplasty
  Arms: XLIMUS DES
Device: Synergy DES Implantation during coronary angioplasty — Synergy DES Implantation during coronary angioplasty
  Arms: Synergy DES

SUMMARY:
The objective of the study is to assess angiographic and clinical performance of Xlimus Drug Eluting Stent (DES) compared to Synergy Bioabsorbable Polymer Everolimus Eluting Stent in patients treated with percutaneous coronary angioplasty

DETAILED DESCRIPTION:
The present clinical investigation is designed as a prospective, multicentre, international, randomized, open label, 2-arm parallel group, trial in patients undergoing Percutaneous Coronary Intervention (PCI) comparing Xlimus DES versus Synergy DES with respect to optical coherence tomography (OCT) derived measures at 6-month Follow Up (FU) and clinical events at 12 months after procedure. A total of 180 patients will be recruited and randomized in the two groups in a 2:1 ratio. After index procedure, patients will be followed up by angiographic follow-up at 6 months and clinical follow-up at 12 months.The primary endpoint will be independently evaluated by the Core-Lab which will be blinded as to group assignment

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18
2. Documented coronary artery disease (CAD): stable or unstable angina, Non-ST segment MI.
3. PCI considered appropriate and feasible
4. Culprit de novo lesion in a native coronary artery with significant stenosis (>50% by visual estimate) eligible for implantation with either study stent (no limitation on the number of treated lesions, vessel and lesion length);
5. Patient provides written informed consent
6. Patient agrees to all required follow-up procedures and visits.
7. Target lesion suitable for PCI with DES diameter between 2.5 and 4.0 mm

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, ticlopidine, sirolimus or its derivatives, everolimus or structurally-related compounds, and/or contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled);
2. Known hypersensitivity to L605 cobalt chromium, 316L stainless steel, platinum, chromium, iron, nickel or molybdenum;
3. Known sensitivity to poly-lactic acid or poly(lactic-co-glycolic acid) polymer;
4. Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrolment into this study and not using adequate contraceptive methods;
5. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions;
6. Previous coronary intervention on target vessel in the 3-months prior to enrollment;
7. Non-cardiac co-morbid conditions with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment);
8. Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period;
9. Previously documented left ventricular ejection fraction (LVEF) <30%;
10. Evident cardiogenic shock before randomization;
11. Patients with left main stem stenosis (>50% by visual estimate);
12. In-stent restenosis;
13. ST-segment elevation MI;
14. Chronic total occlusion/ heavily calcified lesions
15. Culprit lesion to a Saphenous Vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2023-09-02 (Actual)

PRIMARY OUTCOMES:
In-stent neointimal volume | 6-month follow-up
  In-stent neointimal volume at 6-month follow-up, measured with OCT, as assessed by the Core-Lab. Neointimal volume will be calculated in all analyzed cross-sections and volumetric measurements and in stent neointimal volume will be compared in the two groups.

SECONDARY OUTCOMES:
Neointimal area | 6-month follow-up
  Neointimal area calculated at the site of minimal lumen area measured with OCT
Number of Target lesion failure | 12-months follow-up
  composite of Cardiac death, target-vessel Myocardial infarction (MI) and clinically indicated target lesion revascularization (TLR)
Number of patients experiencig Cardiac death | 12-months follow-up
  Any death due to proximate cardiac cause (eg, MI, fatal arrhythmia), unwitnessed death and death of unknown cause, and all procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death
Number of Target-vessel Myocardial infarction | 12-months follow-up
  any MI that, irrespective of the time after the index procedure, is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause. Type of acute MI is classified according to the Joint ESC/ACCF/AHA/ WHF Joint Task Force for the Universal Definition of Myocardial Infarction
Number of Target-lesion revascularization | 12-months follow-up
  repeat revascularization will be defined as any repeat PCI or new coronary artery bypass graft (CABG) surgery within the first year post-PCI
Number of Stent thrombosis | 12-months follow-up
  This is defined according to classification proposed by the Academic Research Consortium
Percentage of Device success at 24 hours | 24 hours
  deployment of the assigned stents without system failure or device-related complication
Percentage of Lesion success at 24 hours | 24 hours
  attainment of <50% residual stenosis of the target lesion using post-PCI
Percentage of Procedural success at 24 hours | 24 hours
  lesion success without the occurrence of major adverse cardiac event (MACE) during the hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Luca Testa, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (4):
- IRCCS Policlinico S. Donato, San Donato Milanese, Milano, Italy
- Spain (3):
  - Hospital Bellvitge, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Testa L, Squillace M, Ventrella N, Moreno R, Jimenez-Valero S, Serra A, Gomez Hospital JA, Bellamoli M, Popolo Rubbio A, Bedogni F. A randomized control trial to assess optical coherence tomography parameters of the Xlimus drug-eluting stent: the XLIMIT trial. Front Cardiovasc Med. 2023 Sep 6;10:1199475. doi: 10.3389/fcvm.2023.1199475. eCollection 2023. PMID 37745092
- [Result] Testa L, Pero G, Bollati M, Casenghi M, Popolo Rubbio A, Cuman M, Moreno R, Serra A, Gomez JA, Bedogni F. XLIMus drug eluting stent: A randomIzed controlled Trial to assess endothelialization. The XLIMIT trial. Int J Cardiol Heart Vasc. 2019 Apr 28;23:100363. doi: 10.1016/j.ijcha.2019.100363. eCollection 2019 Jun. PMID 31061876